CLINICAL TRIAL: NCT06228287
Title: From Great Surgeons to Brilliant Observators, Evolution of Penetrating Neck Trauma in a Single Center Reference in Spain
Acronym: PNT-HMAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Doctor, Hospital del Mar
Other Study IDs: Penetrating neck trauma HMAR
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Penetrating Neck Trauma
Keywords: Penetrating Trauma; Trauma surgery; No zone approach; Non-surgical treatment; Polytrauma
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Penetrating neck trauma ranges from 5 to 10% of trauma patients and its management has been changing in the las 20 years and not all surgeons that attend this patients are trauma surgeons. The aim of the study is to describe the evolution of the management in a referal center and the complications of two periods, with and without a simplified protocol.

DETAILED DESCRIPTION:
Penetrating neck trauma ranges from 5 to 10% of trauma patients and its management has been changing in the las 20 years and not all surgeons that attend this patients are trauma surgeons.

Traditionally, the management was followed by surgical treatment, but the non-therapeutic cervicotomies were ascendent to the 89%, the zone approach was established, following the Monson anatomy zones, with different indications for surgery in every zone, and finally, after the year 2000, started to publish articles on where the injury was not correlated with the zone in about a 23% of the patients.

The aim of the study is to describe the evolution of the management in a referal center and the complications of two periods, with and without a simplified no zone approach protocol.

ELIGIBILITY:
Inclusion Criteria:

* All penetrating trauma patients admitted in the emergency department.

Exclusion Criteria:

* All patients with any other diagnostic different from penetrating trauma
* Blunt trauma patients admitted in the emergency department

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a penetrating trauma in the neck admitted in Hospital del Mar from 2008 to 2022.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Complications | 2008-2022
  The main outcome measure was the total of complications in patients with a penetrating neck trauma assessed by the Clavien-Dindo Classification.
Mortality | 2008-2022
  The second main outcome measure was the total of deaths in patients with a penetrating neck trauma assessed by preventable or non-preventable deaths.
Non-therapeutic cervicotomy | 2008-2022
  The third main outcome measure was the total of non-therapeutic and therapeutic cervitocomies before and after implementing a simplified protocol in patients with a penetrating neck trauma.

SECONDARY OUTCOMES:
Demographyc description | 2008-2022
  Description of the age and gender (Male / Female)
Physiologic description | 2008-2022
  Description of the vitals at arrival (bates per minute, blood pressure)
Wound | 2008-2022
  Description of the wound: bleeding, longitude, number of wounds

CONTACTS AND LOCATIONS:
Overall Officials: Ana María González Castillo, Principal Investigator — Hospital del Mar

IPD SHARING:
Plan to Share IPD: No